CLINICAL TRIAL: NCT03800576
Title: The Influence of Genetic and Clinical Factors on Clinical Outcome of Liver Transplant Patients With Tacrolimus-based Immunosuppression
Brief Title: Clinical Outcome of Liver Transplant Patients With Tacrolimus-based Immunosuppression
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201812015RINC
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2020-01

CONDITIONS: Liver Transplantation
Keywords: tacrolimus; liver transplant; gene polymorphism; immunosuppressant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Genetic polymorphism and numerous clinical factors could influence tacrolimus pharmacokinetics, which led to large inter-and intra-individual variability.Since its narrow therapeutic range,predicting therapeutic outcome and individualized dosage remains to be a challenge. The study's objective is to identify the genetic and clinical factors that can influence clinical outcome in liver transplant.

DETAILED DESCRIPTION:
A great number of studies had found significant correlation between tacrolimus pharmacokinetics and gene polymorphism. However, previous studies on the correlation between genetic factors and clinical outcome were controversial. Furthermore, most studies focused on single genetic polymorphism and clinical outcome, and very limited studies took multiple genetic factors and clinical factors into account.

This is a retrospective study. Eligible patients were those who had signed informed consent for genetic study in previous research projects ( IRB approval number：201512005RINC and 201612023RIND ). The present study will collect laboratory data, concurrent medications, and therapeutic drug monitoring (TDM) data. Patient survival, graft survival, acute rejection and tacrolimus-associated adverse events will be assessed.

ELIGIBILITY:
Eligible patients were those who had signed informed consent for genetic study in our previous research projects.

Inclusion Criteria of the Previous Study:

* patients who underwent living-donor liver transplantation during January 2008 to December 2017
* at the age of 20-65
* with tacrolimus-based immunosuppression after liver transplant for at least 6 months.

Exclusion Criteria of the Previous Study :

* retransplantation
* multi-organ transplantation
* human immunodeficiency virus (HIV) positive.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent living donor liver transplantation (LDLT) during 2008 to 2017 in National Taiwan University Hospital and received tacrolimus-based immunosuppression.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of patients with biopsy proven acute rejection (BPAR) | up to 12 months after liver transplantation
  Incidence of BPAR will be estimated with Kaplan-Meier analysis
Graft survival | up to 9 years after liver transplantation
  incidence of graft loss will be estimated Kaplan-Meier analysis

SECONDARY OUTCOMES:
Number of patients with tacrolimus-associated adverse events | up to 9 years after liver transplantation
  Common adverse events of tacrolimus such as nephrotoxicity, post-transplant diabetes mellitus, hypertension, infection, hyperlipidemia and malignancy.
  * nephrotoxicity：decreased renal function estimated by glomerular filtration rate(GFR) using MDRD 4-Variable Equation
  * Post-transplant diabetes mellitus：defined by diagnosis and the use of antihyperglycemic agents, laboratory data including blood sugar(mg/dL) and hemoglobin A1c (percentage)
  * hypertension：defined by diagnosis and the use of antihypertensive agents, laboratory data including blood pressure(mmHg)
  * infection：defined by diagnosis of infection and the use of antiinfective agents
  * Hyperlipidemia：defined by diagnosis and the use of lipid-lowering agents, laboratory data including LDL (mg/dL), HDL (mg/dL) and total cholesterol (mg/dL)
  * malignancy：incidence of cancer
Patient survival | up to 9 years after liver transplantation
  incidence of death

CONTACTS AND LOCATIONS:
Overall Officials: Rey-Heng Hu, Professor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan